CLINICAL TRIAL: NCT02543021
Title: A Study to Assess the Feasibility and Patient Acceptability of a Randomised, Crossover Design to Compare Virtual vs Conventional Chromoendoscopy for the Detection of Dysplasia in Colitis
Brief Title: Virtual Chromoendoscopy for Colitis Surveillance: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 113398
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Inflammatory Bowel Disease
Keywords: Colitis; Dysplasia; Chromoendoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional chromoendoscopy (Active Comparator): Patients will undergo colitis surveillance colonoscopy with indigo carmine chromoendoscopy (dye spray)
  Interventions: Procedure: Conventional chromoendoscopy
- Virtual chromoendoscopy (Experimental): Patients will undergo colitis surveillance colonoscopy with FICE(TM) virtual chromoendoscopy
  Interventions: Device: Virtual chromoendoscopy

INTERVENTIONS:
Device: Virtual chromoendoscopy — Digital / virtual chromoendoscopy with FICE
  Other Names: Fujinon Intelligent Color Enhancement (FICE)
  Arms: Virtual chromoendoscopy
Procedure: Conventional chromoendoscopy — Conventional chromoendoscopy with indigo carmine dye spray
  Other Names: Indigo carmine dye spray
  Arms: Conventional chromoendoscopy

SUMMARY:
Patients with colitis require regular 'surveillance' colonoscopy as their risk of developing colon cancer is at least 2.5 times that of the general population. However, cancer in colitis develops as flat lesions called dysplasia, that can be easily missed at routine colonoscopy. As a result NICE guidelines for colitis surveillance recommend the use of a technique called chromoendoscopy (CE) in which a water-soluble blue dye is sprayed through the colonoscope to coat and highlight the lining of the bowel, making dysplasia easier to see. Although CE is accepted as best practice for surveillance it is time-consuming, technically difficult and requires expertise to interpret the appearances. For these reasons, its use is not widespread and the vast majority of patients still receive the inferior 'routine' colonoscopy without CE.

New technology means that the video image obtained during colonoscopy can be digitally enhanced and coloured at the press of a button - termed virtual chromoendoscopy (VCE). This could make surveillance colonoscopy shorter, more comfortable and cleaner (resulting in a more 'dignified' experience) as well as cheaper and less technically difficult.

The main objectives to be explored in this feasibility study (and the larger trial) were informed by a PPI meeting, which placed the ability to detect dysplasia at equal importance with the participant's experience of the procedure in terms of speed, comfort and dignity.

This is primarily a feasibility study to assess patient experience, recruitment and retention rates to the investigators' specified trial design, to support the development of a larger crossover trial to compare VCE to CE during surveillance colonoscopy for colitis.

DETAILED DESCRIPTION:
In the recruitment period, 60 patients will be approached when they are invited to attend for scheduled surveillance colonoscopy. Eligible patients (18-75 yrs) who agree to participate will be randomised to undergo CE or VCE as the first procedure. Data will be captured by an Observer using a bespoke Access-based program.

The site and number of any biopsy samples taken will be recorded alongside the Endoscopist's prediction, based on visual appearance, of whether they think the area biopsied is actually dysplasia.

After an agreed interval (no more than 8 weeks, usually 3-6), participants will undergo a second colonoscopy with the second technique, performed by an Endoscopist blinded to the results of the first test, and data captured as before. For each procedure, a questionnaire assessing immediate patient experience will be administered in the Endoscopy department, after the participant has recovered from the procedure. Participants will also be given a second questionnaire assessing their overall experience to take home and complete 48 hours after the procedure, which will be returned by post.

ELIGIBILITY:
Inclusion Criteria:

Any patient eligible for colitis surveillance colonoscopy by British Society of Gastroenterology guidelines:

* Ulcerative pan-proctocolitis or Crohn's colitis of 8 or more years duration
* With or without co-diagnosis of primary sclerosing cholangitis

Exclusion Criteria:

* Inability to provide informed
* Written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Patient adherence to study design - success of recruitment (minimum recruitment of 75%) and retention of patients (minimum target of 75%) | 2 years
  The investigators are evaluating the success of recruitment to the study design with a target minimum recruitment of 75%; The investigators will also evaluate retention of patients within the crossover study design with a minimum target of 75%

SECONDARY OUTCOMES:
Patient experience assessed by validated questionnaire | 2 years
  Patient experience of the procedure in both arms will be compared (intra-individual) by validated questionnaire
Procedure time | 2 years
  The time taken for each procedure will be compared (average)
Miss rate for dysplasia | 2 years
  The miss rate of each technique will be compared
Prediction of histology | 2 years
  The ability of conventional vs virtual chromoendoscopy will be compared to predict eventual histology of targeted biopsies (from which a sensitivity and specificity will be calculated)

CONTACTS AND LOCATIONS:
Overall Officials: Bu'Hussain Hayee, FRCP, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Patient level data will not be shared. Cohort results will form publication/output

REFERENCES:
- [Derived] Pavlidis P, Joshi D, El Sherif Y, Warner B, Gulati S, Alexander J, Cross G, Dew T, Arqoub HA, Devlin J, Heneghan M, Dubois P, Bjarnason I, Powell N, Hayee B. Faecal calprotectin is a surrogate marker of biliary inflammation in primary sclerosing cholangitis associated inflammatory bowel disease. Frontline Gastroenterol. 2022 Mar 18;13(6):497-502. doi: 10.1136/flgastro-2021-102053. eCollection 2022. PMID 36250171